CLINICAL TRIAL: NCT01597765
Title: Effect of Antioxidant Cocktail in Beta-thalassemia/Hb E Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Chiang Mai University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Si 063/2009
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Thalassemia
Keywords: Thalassemia; Oxidative stress; antioxidant cocktail
MeSH Terms: conditions — Thalassemia | interventions — Diarylheptanoids; Acetylcysteine; Deferiprone; Vitamin E; alpha-Tocopherol

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Curcuminoids (Experimental): The administrate curcuminoids is intervention for 30 patients
  Interventions: Drug: curcuminoids, N-acetylcysteine, deferiprone and vitamin E; Drug: Curcuminoids and alpha-tocopherol
- Vitamin E (Experimental): The vitamin E is intervention for 30 patients
  Interventions: Drug: curcuminoids, N-acetylcysteine, deferiprone and vitamin E; Drug: Curcuminoids and alpha-tocopherol

INTERVENTIONS:
Drug: curcuminoids, N-acetylcysteine, deferiprone and vitamin E — receiving curcuminoids 500 mg/day, N-acetylcysteine 200 mg/day deferiprone 50 mg/kg/day and vitamin E 400 IU/day
  Other Names: curcuminoids 500 mg brand name Anti-Ox; N-acetylcysteine 200 mg brand name Mysoven; deferiprone 50 mg/kg/day brand name GPO-L-ONE; vitamin E 400 IU/day brand name Natural
Drug: Curcuminoids and alpha-tocopherol — group 1: receiving curcuminoids 500 mg/day, N-acetylcysteine 200 mg/day and deferiprone 50 mg/kg/day group 2: receiving vitamin E 400 IU/day, N-acetylcysteine 200 mg/day and deferiprone 50 mg/kg/day

SUMMARY:
The purpose of this study is to determine the efficacy of antioxidant cocktails on the alleviation of oxidative stress and iron overload in beta-thalassemia/Hb E patients.

DETAILED DESCRIPTION:
60 cases of beta-thalassemia/Hb E patients. All patients will be diagnosed with hemoglobin typing of beta-thalassemia/Hb E disease and not receive blood transfusion or any treatment at least 3 months prior study. The study will be randomized controlled trial that designed before and after treatment with antioxidant cocktail. The antioxidant cocktail consists of vitamin E 400 IU/day, curcuminoids 500 mg/day, N-acetylcysteine 200 mg/day and deferiprone 50 mg/kg/day. All patients will receive antioxidant cocktail daily for 12 months. The patients will be regularly followed up and analyzed biochemical parameters every two months during treatment and after withdrawal for 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18-50 years
2. hemoglobin level between 6-9 g/dL during screen visit
3. WHO performance status grade 0-2
4. signed in informed consents prior to the study entry.

Exclusion Criteria:

1. receiving iron chelator and blood transfusion.
2. pregnancy or breastfeeding
3. receiving other drugs except folic acid at least 30 days before study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Malonyldiadehyde (MDA) | 1 year after treatment with antioxidant cocktail.
  Lipid peroxidation will be assayed by measuring the formation of malonyldialdehyde (MDA). The formation of MDA on red blood cell will be exposed by hydrogen peroxide. Then, MDA will be extracted by trichloroacetic acid (TCA) and will be reacted with thiobarbituric acid (TBA) in boiling condition to MDA-TBAR complex. This complex will be given pink color and measuring at 532 and 600 nm

CONTACTS AND LOCATIONS:
Overall Officials: Ruchaneekorn Kalpravidh, Assoc. Prof. Dr., Study Chair — Mahidol University
Locations (1):
- Department of Biochemistry , Faculty of Medicine Siriraj Hospital, Mahidol university, Bangkoknoi, Bangkok, Thailand